CLINICAL TRIAL: NCT02707237
Title: Maternal Counseling for Preterm Deliveries, Assessing an Effective Method of Counseling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook County Health (Other Government)
Responsible Party: Principal Investigator, Mopelola Akintorin, MD, Cook County Health
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB 15-226
Record Dates: First submitted 2016-02-08; First posted 2016-03-14 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Pregnancy Preterm; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Verbal counseling (Other): Parents with threatened delivery will receive verbal counseling only
  Interventions: Other: Verbal counseling
- Verbal, pictorial, written counseling (Other): Parents with threatened delivery will receive verbal counseling supplemented with pictorial and written information
  Interventions: Other: Verbal, pictorial, written counseling

INTERVENTIONS:
Other: Verbal counseling — Verbal counseling done by physician
  Arms: Verbal counseling
Other: Verbal, pictorial, written counseling — verbal counseling in addition to gestational age specific written information and pictures will be given to parents
  Arms: Verbal, pictorial, written counseling

SUMMARY:
Providing verbal counseling supplemented with both written and pictorial information then verbal counseling alone is a more effective method of counseling parents with threatened preterm delivery

DETAILED DESCRIPTION:
Progress in the frontiers of neonatology has continually pushed back the limit of viability and significantly improved the survival of extremely preterm infants. An important component of medical management before a preterm delivery is counseling the parents about probabilities of survival and long term complications.

Hypothesis: Preterm counseling is more effective when parents receive verbal counseling supplemented with written and pictorial information then verbal counseling alone.

Methodology: There will be two groups of study (verbal, pictorial and written vs verbal alone). All patients admitted to the L and D department of Stroger hospital between 23 to 34 weeks of gestation with threatened premature delivery will be enrolled in the study. They will be randomly assigned to 1 of 2 groups. After counseling, parents will be asked to complete a 32 point questionnaire to check their knowledge of outcomes of prematurity.

To reach statistically significant results, the investigators will need 40 patients in each group. The study will be done over a period of one year

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 23 to 34 weeks gestation assessed by obstetrician to need counseling

Exclusion Criteria:

* Pregnancies with known life threatening defects considered as non compatible with life.
* Mothers previously admitted and counseled will also be excluded

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2016-03; Primary Completion 2017-10-22 (Actual); Study Completion 2017-10-22 (Actual)

PRIMARY OUTCOMES:
Patient knowledge | one year
  After counseling, patient will answer a 32 point questionnaire and this will be compared across the two groups to see there is any statistical difference between the two groups using SPSS

SECONDARY OUTCOMES:
Maternal anxiety level | one year
  Pre and post counseling administration of 6 item State and Trait anxiety inventory, SPSS software will be used to compute statistical significance

CONTACTS AND LOCATIONS:
Overall Officials: Mopelola Akintorin, MD, Principal Investigator — Cook County Health
Locations (1):
- John H Stroger Jr Hospital of Cook County, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Khashu M, Narayanan M, Bhargava S, Osiovich H. Perinatal outcomes associated with preterm birth at 33 to 36 weeks' gestation: a population-based cohort study. Pediatrics. 2009 Jan;123(1):109-13. doi: 10.1542/peds.2007-3743. PMID 19117868
- [Background] Govande VP, Brasel KJ, Das UG, Koop JI, Lagatta J, Basir MA. Prenatal counseling beyond the threshold of viability. J Perinatol. 2013 May;33(5):358-62. doi: 10.1038/jp.2012.129. Epub 2012 Oct 18. PMID 23079775
- [Background] Blanco F, Suresh G, Howard D, Soll RF. Ensuring accurate knowledge of prematurity outcomes for prenatal counseling. Pediatrics. 2005 Apr;115(4):e478-87. doi: 10.1542/peds.2004-1417. PMID 15805351
- [Background] Muthusamy AD, Leuthner S, Gaebler-Uhing C, Hoffmann RG, Li SH, Basir MA. Supplemental written information improves prenatal counseling: a randomized trial. Pediatrics. 2012 May;129(5):e1269-74. doi: 10.1542/peds.2011-1702. Epub 2012 Apr 9. PMID 22492766
- [Derived] Budhani S, Akintorin M, Soyemi K, Fogg L, Arlandson M, Kumar R. Maternal counseling for preterm deliveries, assessing an effective method of counseling: A randomized trial. PLoS One. 2025 Apr 9;20(4):e0294168. doi: 10.1371/journal.pone.0294168. eCollection 2025. PMID 40203068